CLINICAL TRIAL: NCT01767259
Title: Pharmacokinetic Interactions of Valsartan and Hydrochlorothiazide: An Open-Label, Randomized, Four-Period Crossover Study in Healthy Egyptian Male Volunteers
Brief Title: Pharmacokinetic Interactions of Valsartan and Hydrochlorothiazide
Acronym: PKVH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Sally Helmy, PhD, CPHQ, Lecturer of Pharmaceutics, Faculty of Pharmacy, Damanhour University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PPT1
Record Dates: First submitted 2013-01-08; First posted 2013-01-14 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Normotensive Participants
Keywords: Fixed dose combination; Pharmacokinetics; Valsartan; Hydrochlorothiazide
MeSH Terms: interventions — Valsartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Valsartan 160 mg alone (Other): Valsartan alone
  Interventions: Drug: Valsartan
- Hydrochlorothiazide 12.5 mg alone (Other): Hydrochlorothiazide alone
  Interventions: Drug: Hydrochlorothiazide
- Valsartan160 mg + Hydrochlorothiazide12.5 mg (Other): Concomitant administration of valsartan 160 mg + Hydrochlorothiazide 12.5 mg
  Interventions: Drug: Valsartan/Hydrochlorothiazide
- Valsartan / Hydrochlorothiazide 160 mg/12.5mg (Other): Fixed dose combination of valsartan 160 mg + Hydrochlorothiazide 12.5 mg
  Interventions: Drug: Valsartan/Hydrochlorothiazide

INTERVENTIONS:
Drug: Valsartan/Hydrochlorothiazide — Co-administration or fixed dose combination
  Other Names: Fixed dose combination; Pharmacokinetic interaction
  Arms: Valsartan / Hydrochlorothiazide 160 mg/12.5mg; Valsartan160 mg + Hydrochlorothiazide12.5 mg
Drug: Valsartan — Valsartan alone
  Arms: Valsartan 160 mg alone
Drug: Hydrochlorothiazide — Hydrochlorothiazide alone
  Arms: Hydrochlorothiazide 12.5 mg alone

SUMMARY:
This study was conducted to compare the rate and extent of absorption of valsartan and hydrochlorothiazide following oral administration as a fixed dose combination tablet and concomitant administration of the individual drugs under fasting conditions in healthy Egyptian subjects. The study was extended to investigate any potential reaction between VAL and HCT.

DETAILED DESCRIPTION:
This study comprised 2 separate parts, I and II; each was a single-dose, open-label, 4-crossover periods separated by a 2 weeks washout, and 4-Treatments. Part I consisted of Treatments A (VAL 160 mg alone), B (HCT 12.5 mg alone), C (VAL 160 mg + HCT 12.5 mg) and D (VAL / HCT 160 mg/12.5mg) and Part II consisted of Treatments E (VAL 320 mg alone), F (HCT 25 mg alone), G (VAL 320 mg + HCT 25 mg) and H (VAL / HCT 320 mg/25 mg). Blood samples were collected up to 48 hours postdose and plasma was analyzed for VAL and HCT concentrations using HPLC. The pharmacokinetic properties of each drug after co-administration of VAL and HCT were compared with those of each drug administered alone.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and not more than 45 healthy male volunteers
* Actual weight no more than ± 30% from ideal body weight based on sex, height, and body frame
* Who had passed all the screening parameters
* Free of any drug exposure known to interfere with the pharmacokinetics or assay of fexofenadine for at least 10 days prior to the study
* Who had to be able to communicate effectively with study personnel, be literate, and able to give consent.

Exclusion Criteria:

* A clinically significant abnormal physical exam, medical history, or laboratory studies
* If they showed a sitting SBP of >140 or <100 mmHg, DBP > 90 or <60mm Hg, or a pulse rate of > 95 or < 50 beats/min at screening
* A history of serious intolerance, allergy, or sensitivity to fexofenadine
* The use of any prescription drug within the previous month or use of any over-the-counter medication (with the exception of acetaminophen) within the past 14 days
* A history of blood dyscrasias
* A history of alcohol or drug abuse within the past year
* Donation of blood during the 8 weeks prior to the study or plans to donate blood during or within 8 weeks of completing the study
* Unable to tolerate vein puncture and multiple blood samplings
* Any surgical/medical condition that might alter drug absorption, distribution, metabolism, or excretion
* Cannot follow instructions, in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tolerability | Participants will be followed for the duration of study, an expected average of 6 weeks.
  Tolerability was assessed based on changes in vital signs (temperature, blood pressure, pulse, and heart rate), measured before dosing in each period and approximately every 4 hours thereafter, and laboratory tests (hematology, biochemistry, liver function, and urinalysis), and performed at baseline and at the end of the study. In addition, a physician questioned volunteers about any adverse events occurring during the study, addressed them as necessary, and recorded them on the appropriate form. This physician was not blinded to treatment, but had no involvement in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Helmy, PhD, CPHQ, Principal Investigator — Pharmaceutics Department, Faculty of Pharmacy, Damanhour University, Damanhour, Egypt
Locations (1):
- Pharmaceutics Department, Faculty of Pharmacy, Damanhour University, Damanhur, Egypt